CLINICAL TRIAL: NCT04899934
Title: Multi-Site Feasibility Evaluation of Crisis Stabilization Units Across Three Jurisdictions With High Opioid Use Disorders and a Proposed Follow-Up RCT
Brief Title: Feasibility of Mobile and Technology Assisted Aftercare Services for Crisis Stabilization Units
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Carrie Pettus-Davis, associate professor; founder and executive director Institute of Justice Research & Development, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00001570; 19-02811 (Other Grant/Funding Number: Arnold Venture)
Record Dates: First submitted 2021-04-30; First posted 2021-05-25 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Substance Abuse; Criminal Behavior; Mental Disorder
Keywords: crisis stabilization; psychological well-being; law enforcement; mental health treatment; substance use disorder treatment
MeSH Terms: conditions — Substance-Related Disorders; Criminal Behavior; Mental Disorders; Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: A total of 24 adults releasing to one of the three participating counties in Florida will be randomly assigned to participate in the mobile and technology assisted aftercare or a treatment-as-usual (TAU) control group. Participants assigned to the treatment-as-usual control group will remain eligible to participate in all agency specific services offered to persons discharging the CSU as well as, any community resources they normally would have access to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile and technology assisted aftercare (Experimental): participants randomized to this condition will receive up to 26 sessions with a community support specialist aftercare provider and 6 months of access to behavioral health mobile applications.
  Interventions: Behavioral: mobile and technology assisted aftercare
- Treatment as usual (TAU) (Active Comparator): Participants randomized to this condition receive standard treatment services available to persons discharging from a CSU.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: mobile and technology assisted aftercare — The mobile and technology assisted aftercare consists of mobile mental health professionals who travel to participants to provide mental health services including counseling, navigation of community referrals, motivational interviewing, solution focused therapy, psycho-education, and social support. Participants randomized to this condition will also receive 24/7 access to evidence-based behavioral health mobile applications that are recommended based on the participant's diagnostic status, learning style, and goals. Frequency of app use is up to the participant's discretion. However, during weekly aftercare sessions, the CSS may assist the participant with creation of an app use schedule that is realistic for the participant's needs and treatment goals.
  Arms: Mobile and technology assisted aftercare
Other: Treatment as usual — Treatment as usual services include a personalized discharge plan, a follow up appointment within a month of discharge for evaluation and connection to other agency services if applicable. Some of these services may include outpatient counseling for behavioral and emotional problems, psychiatric services, group therapy, case management, rehabilitation services, homeless recovery services, employment services, medication-assisted treatment, group-based team building activities, primary care clinic, and forensic services. Individuals may also receive ancillary referrals for applicable healthcare services, access to residential and outpatient substance abuse treatment services, and access to a tablet.
  Arms: Treatment as usual (TAU)

SUMMARY:
In this study investigators are examining the feasibility and acceptability of an expanded and technology-assisted aftercare program with persons released from a crisis stabilization unit (CSU) who were brought to the CSU by choice of law enforcement. Investigators are assessing the critical elements of CSUs, examining the feasibility and acceptability of pairing mobile and technology-assisted aftercare to improve treatment access and retention; and developing a study protocol to be used in a future multisite randomized controlled trial (RCT).

Crisis stabilization units provide law enforcement officers an alternative to jail for individuals experiencing a substance use or mental health disorder crisis contributing to criminalized behavior. This study is designed to assist with the diversion of individuals toward treatment and away from subsequent contact with law enforcement through piloting mobile and technology assisted aftercare services to persons released from a CSU. One of the largest barriers to the effectiveness of CSUs is retaining the individual in treatment after discharge. Logistical factors including transportation, stable housing, and long waitlists for community-based treatment decrease treatment access. These factors may also be complicated by an individual's understanding of the importance of remaining in treatment as well as their motivation to continue. To overcome these barriers and enhance the impact of CSUs, investigators are developing an expanded model which includes mobile and technology-assisted modalities that address psychological, behavioral, and medication-assisted treatment.

DETAILED DESCRIPTION:
This study is a mixed methods design, combining a randomized controlled trial and qualitative interviews into the feasibility of the pilot program, mobile and technology assisted aftercare. The randomized controlled trial consists of a 1:1 comparison of the pilot CSU aftercare services and the treatment as usual (TAU) services for persons releasing from a CSU.

Participants (n=24) are recruited into the study prior to their discharge from a CSU. Research team members are alerted of potential eligible participants who meet study criteria and are soon-to-be discharged by CSU staff. At this point, research team members approach the eligible participants to conduct the recruitment and consent process. Due to the short length of stay in a CSU, the research team does one-to-one randomization and pre-randomize of the pool of participants prior to recruitment. For example, the pre-randomization may results in Tx Tx Ctrl Tx Ctrl Ctrl assignments for each sequential enrollment in the study. Or it may result in a different pattern Ctrl Txt Ctrl, etc. Participants are notified of their randomization status at the end of the consent and baseline data collection interview.

The pilot program of mobile and technology assisted aftercare service connects participants with a Community Support Specialist (CSS) who provides mobile aftercare (i.e., meet the client in their homes or other community settings) up to once a week for 6 months. Participants also have 24/7 access to behavioral health mobile applications on a smart phone. Mobile apps recommended to participants include, moodtools-depression aid, virtual hope box, recovery path, and intellicare hub. All mobile apps have undergone one or a combination of RCTs, clinical trials, and/or developed with mental health professionals.

Data is collected through participant interviews and collection of health and administrative records from agency collaborators. Participants will complete a total of 4 interviews over a period of 6 months. Baseline interviews will be conducted at study enrollment. Time 1 (T1) interviews will be conducted 2 weeks post-discharge from the CSU. Time 2 (T2) interviews will be conducted 3 months post-discharge from CSU. Time 3 (T3) will be conducted 6 months post-discharge from the CSU. The investigators are monitoring trends in participants during their participation in the pilot program and all consented participants for the treatment and control groups will complete a series of interviews. The assessed trends include readmission to a CSU, employment stability, financial stability, criminal justice involvement, perception of social support, use of acute and long-term services, and multiple psychosocial measures listed below.

Data assessing the feasibility and acceptability of the mobile and technology-assisted aftercare is also assessed through qualitative interviews and focus groups with our community mental health partner. This qualitative data will be used to create a protocol for CSU aftercare that can respond to diverse jurisdictional characteristics leading to CSU aftercare services that are feasible and scalable.

ELIGIBILITY:
Inclusion Criteria:

* brought to Meridian Behavioral Health CSU by the choice of law enforcement
* over 18 years of age
* self-report to be residing in Alachua, Columbia, or Levy county for at least 6 months following their discharge from the CSU.
* conversational in English
* being able to cognitively consent

Exclusion Criteria:

* younger than 18 years old
* not cognitively able to consent
* not conversational in English
* not releasing from the CSU to Alachua, Columbia, or Levy County, Florida
* not brought to the CSU by choice of law enforcement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited | up to 6 months
  Number of eligible participant who agree to participate out of total number of eligible participants
Retention of participants | up to 6 months
  Retention of participants is tracked by the number of recruited participants who complete the intervention
Number of intervention sessions completed | up to 6 months
  Number of intervention sessions completed is tracked by the number of sessions participants complete over 6 months

SECONDARY OUTCOMES:
Change in arrest rates | up to 6 months
  Change in arrest rates will be tracked by the number of arrests participants incur over a 6-month period beginning at baseline
Frequency of acute service use | up to 6 months
  Frequency of acute service use is tracked by the number of acute services participants partake in over a 6-month period beginning at baseline
Frequency of long-term treatment use | up to 6 months
  Frequency of long-term treatment use if tracked by the number of long-term treatment services participants partake in over a 6-month period beginning at baseline
Admission into a crisis stabilization unit | up to 6 months
  Admission into a crisis stabilization unit is tracked by the number of times a participant is admitted into a crisis stabilization unit over a 6-month period beginning at baseline
Acceptability of intervention specific aftercare services | up to 12 months
  Acceptability of intervention specific aftercare services is assessed through qualitative interviews with mental health stakeholders and CSU staff

OTHER OUTCOMES:
Change in law breaking behavior | 2 weeks post-release
  Change in law breaking behavior is tracked by a dichotomous "yes" or "no" survey in which participants are asked about law breaking behavior including if they had contact with police, if they participated in an activity that would have resulted in legal consequence had they been caught, or if they failed to pay child support.
Change in law breaking behavior | 3 months post-release
  Change in law breaking behavior is tracked by a dichotomous "yes" or "no" survey in which participants are asked about law breaking behavior including if they had contact with police, if they participated in an activity that would have resulted in legal consequence had they been caught, or if they failed to pay child support.
Change in law breaking behavior | 6 months post-release
  Change in law breaking behavior is tracked by a dichotomous "yes" or "no" survey in which participants are asked about law breaking behavior including if they had contact with police, if they participated in an activity that would have resulted in legal consequence had they been caught, or if they failed to pay child support.
Change in financial stability | 2 weeks post-release
  Financial stability was defined as an ability to pay for one's bills, basic needs, and a potential unexpected expense without difficultly. Various intensity scales (0 = none/never to 5 = all of the time) and dichotomous "yes" "no" questions on an 8 question survey capture the participant's financial stability. The lower the score the greater the financial stability.
Change in financial stability | 3 months post-release
  Financial stability was defined as an ability to pay for one's bills, basic needs, and a potential unexpected expense without difficultly. Various intensity scales (0 = none/never to 5 = all of the time) and dichotomous "yes" "no" questions on an 8 question survey capture the participant's financial stability.The lower the score the greater the financial stability.
Change in financial stability | 6 months post-release
  Financial stability was defined as an ability to pay for one's bills, basic needs, and a potential unexpected expense without difficultly. Various intensity scales (0 = none/never to 5 = all of the time) and dichotomous "yes" "no" questions on an 8 question survey capture the participant's financial stability.The lower the score the greater the financial stability.
Change in perception of social support | 2 weeks post release
  Perception of social support was defined as the number of socially supportive characteristics (such as being someone they count on, are emotionally close with, can be themselves with, feel relaxed around, and feel valued by) present in 3 people in the participant's "social network." Participants are asked an identical set of 23 questions about these 3 people to capture their perception of the presence of socially supportive characteristics. Various intensity scales are used where (0= the least perception or never to 5 = the most perception of support or always). Dichotomous 'yes" and "no" questions are also used to capture participant's perception of the social support characteristics within their social network. The higher the score the greater the perception of social support.
Change in perception of social support | 3 months post release
  Perception of social support was defined as the number of socially supportive characteristics (such as being someone they count on, are emotionally close with, can be themselves with, feel relaxed around, and feel valued by) present in 3 people in the participant's "social network." Participants are asked an identical set of 23 questions about these 3 people to capture their perception of the presence of socially supportive characteristics. Various intensity scales are used where (0= the least perception or never to 5 = the most perception of support or always). Dichotomous 'yes" and "no" questions are also used to capture participant's perception of the social support characteristics within their social network. The higher the score the greater the perception of social support.
Change in perception of social support | 6 months post release
  Perception of social support was defined as the number of socially supportive characteristics (such as being someone they count on, are emotionally close with, can be themselves with, feel relaxed around, and feel valued by) present in 3 people in the participant's "social network." Participants are asked an identical set of 23 questions about these 3 people to capture their perception of the presence of socially supportive characteristics. Various intensity scales are used where (0= the least perception or never to 5 = the most perception of support or always). Dichotomous 'yes" and "no" questions are also used to capture participant's perception of the social support characteristics within their social network.The higher the score the greater the perception of social support.
Change in psychological well-being | 2 weeks post release
  Psychological well-being is a complex combination of various psychological and personality characteristics and may be marked by the absence of mental and emotional disturbances including feelings of hopelessness, loneliness, anxiety, paranoia, or fear. psychological well-being is measured by the Brief Symptom Inventory, 53 items with a 6 question sub-scale of psychological symptoms were a respondent characterizes the intensity of mental and emotional disturbances (0= "not at all" to 4 - "extremely"). The higher the score the less psychological well-being present.
Change in psychological well-being | 3 months post release
  Psychological well-being is a complex combination fo various psychological and personality characteristics and may be marked by the absence of mental and emotional disturbances including feelings of hopelessness, loneliness, anxiety, paranoia, or fear. psychological well-being is measured by the Brief Symptom Inventory, 53 items with a 6 question sub-scale of psychological symptoms were a respondent characterizes the intensity of mental and emotional disturbances (0= "not at all" to 4 - "extremely"). The higher the score the less psychological well-being present.
Change in psychological well-being | 6 months post release
  Psychological well-being is a complex combination of various psychological and personality characteristics and may be marked by the absence of mental and emotional disturbances including feelings of hopelessness, loneliness, anxiety, paranoia, or fear. psychological well-being is measured by the Brief Symptom Inventory, 53 items with a 6 question sub-scale of psychological symptoms were a respondent characterizes the intensity of mental and emotional disturbances (0= "not at all" to 4 - "extremely"). The higher the score the less psychological well-being present.
Change in employment stability | 2 weeks post release
  Employment stability is captured with an 11-item questionnaire that uses a combination of dichotomous "yes" or "no" questions and open-ended short answer questions to assess employment stability. Employment stability is defined through employment status, employment duration, employment history, and sources of income.
Change in employment stability | 3 months post release
  Employment stability is captured with an 11-item questionnaire that uses a combination of dichotomous "yes" or "no" questions and open-ended short answer questions to assess employment stability. Employment stability is defined through employment status, employment duration, employment history, and sources of income.
Change in employment stability | 6 months post release
  Employment stability is captured with an 11-item questionnaire that uses a combination of dichotomous "yes" or "no" questions and open-ended short answer questions to assess employment stability. Employment stability is defined through employment status, employment duration, employment history, and sources of income.
Change in coping self-efficacy | 2 weeks post release
  Self-efficacy is a cognitive mechanism based on expectation or beliefs about one's ability to perform actions necessary to produce a given effect. The 28 item Brief Cope index assess coping self-efficacy and confidence coping with stress using an intensity scale (1= "never" to 4 = "always"). The higher the score the greater the coping self-efficacy.
Change in coping self-efficacy | 3 months post release
  Self-efficacy is a cognitive mechanism based on expectation or beliefs about one's ability to perform actions necessary to produce a given effect. The 28 item Brief Cope index assess coping self-efficacy and confidence coping with stress using an intensity scale (1= "never" to 4 = "always"). The higher the score the greater the coping self-efficacy.
Change in coping self-efficacy | 6 months post release
  Self-efficacy is a cognitive mechanism based on expectation or beliefs about one's ability to perform actions necessary to produce a given effect. The 28 item Brief Cope index assess coping self-efficacy and confidence coping with stress using an intensity scale (1= "never" to 4 = "always"). The higher the score the greater the coping self-efficacy.
Change in psychological trauma | 2 weeks post release
  Psychological trauma is identified as an emotionally painful, shocking, stressful, and sometimes life-threatening experience. The 25-item Trauma History Questionnaire assess the occurrence of psychological trauma over the lifetime with dichotomous "yes" or "no" questions, then respondents are asked to self-report the age they were at the time of the incident and frequency the trauma occurred.
Change in psychological trauma | 3 months post release
  Psychological trauma is identified as an emotionally painful, shocking, stressful, and sometimes life-threatening experience. The 25-item Trauma History Questionnaire assess the occurrence of psychological trauma over the previous 3 months with dichotomous "yes" or "no" questions, then respondents are asked to self-report the age they were at the time of the incident and frequency the trauma occurred.
Change in psychological trauma | 6 months post release
  Psychological trauma is identified as an emotionally painful, shocking, stressful, and sometimes life-threatening experience. The 25-item Trauma History Questionnaire assess the occurrence of psychological trauma over the previous 3 months with dichotomous "yes" or "no" questions, then respondents are asked to self-report the age they were at the time of the incident and frequency the trauma occurred.
Change in therapeutic alliance | 2 weeks post release
  Therapeutic alliance is identified as a relationship factor in counseling that includes three dimensions: goal consensus between counselor and client, collaboration on counseling-related tasks, and emotional bonding. Therapeutic alliance is assessed by the California Group Psychotherapy Alliance Scale, with 24 items on an intensity scale with 1 indicating "not at all" and 7 indicating "very much so." The lower the score the greater the therapeutic alliance.
Change in therapeutic alliance | 3 months post release
  Therapeutic alliance is identified as a relationship factor in counseling that includes three dimensions: goal consensus between counselor and client, collaboration on counseling-related tasks, and emotional bonding. Therapeutic alliance is assessed by the California Group Psychotherapy Alliance Scale, with 24 items on an intensity scale with 1 indicating "not at all" and 7 indicating "very much so." The lower the score the greater the therapeutic alliance.
Change in therapeutic alliance | 6 months post release
  Therapeutic alliance is identified as a relationship factor in counseling that includes three dimensions: goal consensus between counselor and client, collaboration on counseling-related tasks, and emotional bonding. Therapeutic alliance is assessed by the California Group Psychotherapy Alliance Scale, with 24 items on an intensity scale with 1 indicating "not at all" and 7 indicating "very much so." The lower the score the greater the therapeutic alliance.
Change in technology use | 2 weeks post release
  Technology use is a 4 item qualitative questionnaire that assess respondents frequency of use, likes, and dislikes, of recommended behavioral health mobile applications.
Change in technology use | 3 months post release
  Technology use is a 4 item qualitative questionnaire that assess respondents frequency of use, likes, and dislikes, of recommended behavioral health mobile applications.
Change in technology use | 6 months post release
  Technology use is a 4 item qualitative questionnaire that assess respondents frequency of use, likes, and dislikes, of recommended behavioral health mobile applications.
Perception of police interaction | baseline
  Police interaction is defined as any physical contact with police and is assessed with the Police Contact Interaction Survey, a 30-item questionnaire with various intensity scales ranging from 1-4 where 1 = less satisfied and 4 = more satisfied with the police interaction. The survey also includes dichotomous "yes" or "no" questions where respondents identify if the police officer did a certain action. Respondents are asked to consider the police interaction that resulted in them being brought to the CSU.
Perception of police interaction | 2 weeks post release
  Police interaction is defined as any physical contact with police and is assessed with the Police Contact Interaction Survey, a 30-item questionnaire with various intensity scales ranging from 1-4 where 1 = less satisfied and 4 = more satisfied with the police interaction. The survey also includes dichotomous "yes" or "no" questions where respondents identify if the police officer did a certain action. Respondents are asked to consider any police interaction occurring within the last 2 weeks.
Perception of police interaction | 3 months post release
  Police interaction is defined as any physical contact with police and is assessed with the Police Contact Interaction Survey, a 30-item questionnaire with various intensity scales ranging from 1-4 where 1 = less satisfied and 4 = more satisfied with the police interaction. The survey also includes dichotomous "yes" or "no" questions where respondents identify if the police officer did a certain action. Respondents are asked to consider any police interaction occurring within the last 3 months.
Perception of police interaction | 6 months post release
  Police interaction is defined as any physical contact with police and is assessed with the Police Contact Interaction Survey, a 30-item questionnaire with various intensity scales ranging from 1-4 where 1 = less satisfied and 4 = more satisfied with the police interaction. The survey also includes dichotomous "yes" or "no" questions where respondents identify if the police officer did a certain action. Respondents are asked to consider any police interaction occurring within the last 3 months.
Change in hope self-efficacy | 2 weeks post release
  Self-efficacy is a cognitive mechanism based on expectation or beliefs about one's ability to perform actions necessary to produce a given effect. The Hearth Hope Index assess hope self-efficacy and a respondent's outlook on life with a 12-item questionnaire where responses are rated on an intensity scale 1-4 (1= "strongly disagree" to 4= "strongly agree"). The higher the score the more hope.
Change in hope self-efficacy | 3 months post release
  Self-efficacy is a cognitive mechanism based on expectation or beliefs about one's ability to perform actions necessary to produce a given effect. The Hearth Hope Index assess hope self-efficacy and a respondent's outlook on life with a 12-item questionnaire where responses are rated on an intensity scale 1-4 (1= "strongly disagree" to 4= "strongly agree"). The higher the score the more hope.
Change in hope self-efficacy | 6 months post release
  Self-efficacy is a cognitive mechanism based on expectation or beliefs about one's ability to perform actions necessary to produce a given effect. The Hearth Hope Index assess hope self-efficacy and a respondent's outlook on life with a 12-item questionnaire where responses are rated on an intensity scale 1-4 (1= "strongly disagree" to 4= "strongly agree"). The higher the score the more hope.
Change in employment aspiration | 2 weeks post release
  Employment aspiration was defined as a desire and willingness to adjust one's employment situation. The Employment Education Aspiration Satisfaction assess education aspiration with a 13-item questionnaire where responses are rated on an intensity scale 1-4 (1= "strongly disagree" to 4= "strongly agree"). The higher the score the more employment aspiration.
Change in employment aspiration | 3 months post release
  Employment aspiration was defined as a desire and willingness to adjust one's employment situation. The Employment Education Aspiration Satisfaction assess education aspiration with a 13-item questionnaire where responses are rated on an intensity scale 1-4 (1= "strongly disagree" to 4= "strongly agree"). The higher the score the more employment aspiration.
Change in employment aspiration | 6 months post release
  Employment aspiration was defined as a desire and willingness to adjust one's employment situation. The Employment Education Aspiration Satisfaction assess education aspiration with a 13-item questionnaire where responses are rated on an intensity scale 1-4 (1= "strongly disagree" to 4= "strongly agree"). The higher the score the more employment aspiration.
Change in education aspiration | 2 weeks post release
  Education aspiration was defined as a desire and willingness to increase one's education. The Employment Education Aspiration Satisfaction assess education aspiration with a 13-item questionnaire where responses are rated on an intensity scale 1-4 (1= "strongly disagree" to 4= "strongly agree"). The higher the score the more education aspiration.
Change in education aspiration | 3 months post release
  Education aspiration was defined as a desire and willingness to increase one's education. The Employment Education Aspiration Satisfaction assess education aspiration with a 13-item questionnaire where responses are rated on an intensity scale 1-4 (1= "strongly disagree" to 4= "strongly agree"). The higher the score the more education aspiration.
Change in education aspiration | 6 months post release
  Education aspiration was defined as a desire and willingness to increase one's education. The Employment Education Aspiration Satisfaction assess education aspiration with a 13-item questionnaire where responses are rated on an intensity scale 1-4 (1= "strongly disagree" to 4= "strongly agree"). The higher the score the more education aspiration.
Change in need for community services | 2 weeks post release
  Change in need for community services is tracked using a service assessment questionnaire that captures the perceived need and use of services in areas of cognitive, housing, relationships, health, education, job readiness, substance abuse, mental health, and life skills. The service assessment questionnaire include dichotomous "yes" "no" questions, a continuum where respondents report "how many times" they received a service, and asks participants why they could not receive a service they perceived themself as needing.
Change in need for community services | 3 months post release
  Change in need for community services is tracked using a service assessment questionnaire that captures the perceived need and use of services in areas of cognitive, housing, relationships, health, education, job readiness, substance abuse, mental health, and life skills. The service assessment questionnaire include dichotomous "yes" "no" questions, a continuum where respondents report "how many times" they received a service, and asks participants why they could not receive a service they perceived themself as needing.
Change in need for community services | 6 months post release
  Change in need for community services is tracked using a service assessment questionnaire that captures the perceived need and use of services in areas of cognitive, housing, relationships, health, education, job readiness, substance abuse, mental health, and life skills. The service assessment questionnaire include dichotomous "yes" "no" questions, a continuum where respondents report "how many times" they received a service, and asks participants why they could not receive a service they perceived themself as needing.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Pettus, PHD, Principal Investigator — Florida State University College of Social Work, Institute for Justice Research and Development
Locations (1):
- Institute for Justice Research and Development, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pettus C, Fulmer R, Pederson SD, Eikenberry J. Study protocol paper for the multi-site feasibility evaluation of mobile and technology-assisted aftercare services for crisis stabilization units. Pilot Feasibility Stud. 2023 Jul 31;9(1):135. doi: 10.1186/s40814-023-01361-8. PMID 37525253